CLINICAL TRIAL: NCT03999788
Title: Clinical Relevance of miR-142-3p as Potential Biomarker of Synaptopathy in Multiple Sclerosis
Brief Title: miR-142-3p as Potential Biomarker of Synaptopathy in MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Haed of Neurology Unit, Neuromed IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: miR-142-3p_MSSynPathyBiomarker; RF-2018-12366144 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2019-06-21; First posted 2019-06-27 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis; Spasticity
Keywords: microRNA; Multiple Sclerosis; synaptopathy; lower limb spasticity; transcranial magnetic stimulation; repetitive TMS stimulation protocol; GLAST/EAAT1; single nucleotide polymorphisms; Intermittent theta burst stimulation (iTBS)
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multiple sclerosis patients (Experimental): lumbar puncture, microRNAs quantification in CSF samples, SNPs analysis in blood samples
  Interventions: Procedure: lumbar puncture and blood withdrawal
- control subjects (Experimental): lumbar puncture, microRNAs quantification in CSF samples, SNPs analysis in blood samples
  Interventions: Procedure: lumbar puncture and blood withdrawal
- multiple sclerosis patients with spasticity and selected SNPs (Experimental): iTBS therapeutic protocol
  Interventions: Procedure: Intermittent theta burst stimulation (iTBS) therapeutic protocol for spasticity

INTERVENTIONS:
Procedure: lumbar puncture and blood withdrawal — lumbar puncture performed to detect OCB for diagnostic purposes and blood withdrawal for SNP screening
  Arms: control subjects; multiple sclerosis patients
Procedure: Intermittent theta burst stimulation (iTBS) therapeutic protocol for spasticity — iTBS will be delivered over the scalp site corresponding to the leg area of primary motor cortex contralateral to the affected limb. The active motor threshold (AMT) will be defined as the minimum stimulation intensity required to evoke a liminal motor potential from the Soleus muscle during voluntary contraction. The stimulation intensity will be about 80% of AMT. The iTBS stimulation protocol consists of 10 bursts, each burst composed of three stimuli at 50 Hz, repeated at a theta frequency of 5 Hz every 10 s for a total of 600 stimuli (200 s). If no MEP will be detectable from the contralateral leg, the site of stimulation will be determined as symmetrical to the motor hot spot. If no MEP will be detectable even from the contralateral leg the coil will be held tangentially to the scalp with its centre placed 1 cm ahead and 1 cm lateral from CZ (10-20 EEG system). In these cases, stimulation intensity will be set to 50% of the maximum stimulator output.
  Arms: multiple sclerosis patients with spasticity and selected SNPs

SUMMARY:
Inflammatory synaptopathy is a prominent pathogenic mechanism in multiple sclerosis (MS) and in its mouse model, which can cause excitotoxic damage by long-lasting excessive synaptic excitation and, consequentially, drives disease progression by leading to motor and cognitive deficits. As synaptopathy occurs early during the disease course and is potentially reversible, it represents an appealing therapeutic target in MS.

Although reliable biomarkers of MS synaptopathy are still missing, recent researches highlighted miR-142-3p as a possible candidate. Indeed, miR-142-3p has been described to promote the IL-1beta-dependent synaptopathy by downregulating GLAST/EAAT1, a crucial glial transporter involved in glutamate homeostasis. Furthermore, mir-142-3p has been suggested as a putative negative MS prognostic factor and a target of current MS disease modifying therapies.

The hypothesis of this study is that miR-142-3p represents a good biomarker for excitotoxic synaptopathy to predict MS course, and, possibly, treatment efficacy at individual level, including both pharmacological strategies and non-pharmacological interventions, like therapeutic transcranial magnetic stimulation (TMS) to ameliorate MS spasticity. To this aim, the role of miR-142-3p in MS synaptopathy, its potential impact on the efficacy of disease-modifying treatments currently used in MS therapy as well as the influence of genetic variants (SNPs) of miR-142-3p and GLAST/EAAT1 coding genes on the responsiveness to therapeutic TMS, will be further investigated in the study. By validating miR-142-3p as potential biomarker of synaptopathy, it is expect to improve MS prognosis and personalized therapies.

Patients with MS, who will undergo neurological assessment, conventional brain MRI scan, and CSF and blood withdrawal for diagnostic and clinical reasons at the Neurology Unit of IRCCS INM-Neuromed will be enrolled in the study. Neurophysiological, biochemical and genetic parameters together with lower limb spasticity will be evaluated. Subjects, who will undergo blood sampling and/or lumbar puncture for clinical suspicions, later on not confirmed, will be recruited as control group.

A subgroup of MS patients showing lower limb spasticity will be included in a two-week repetitive TMS stimulation protocol (iTBS) to correlate the patient responsiveness to this non-pharmacological treatment with MS-significant SNPs of both miR-142-3p and GLAST/EAAT1 coding genes.

DETAILED DESCRIPTION:
In the last decade, structural and functional synaptic alterations, collectively known as synaptopathy, have come up as a determinant pathological process contributing to the neurodegenerative damage in multiple sclerosis (MS) and its mouse model, the experimental autoimmune encephalomyelitis (EAE). Since synaptic alteration and loss are reversible, unlike loss of neurons, an early detection could permit a precocious clinical intervention with potentially better therapeutic outcomes but reliable biomarkers are not available yet.

MicroRNAs (miRs) circulating in the cerebrospinal fluids (CSF) are good candidates as possible sensitive biomarkers for MS synaptopathy-driven disease progression. They represent a new class of modulators of gene expression with stable presence in the body fluids and with a critical role in many physiological and pathological processes, especially in the central nervous system. Accordingly, it has been recently demonstrated that miR-142-3p is a crucial component in a detrimental regulatory axis of EAE/MS excitotoxic synaptic dysfunctions, by reducing the level of the glial glutamate aspartate transporter/excitatory amino acid transporter 1 (GLAST/EAAT1) protein. Moreover, miR-142-3p levels are increased in both EAE brains and CSFs of patients with relapsing-remitting MS (RRMS) and correlate with disease progression. Preliminary data also reveal that miR-142-3p is direct target of different pharmacological treatments for MS, while the action of non-pharmacological treatments, as therapeutic transcranial magnetic stimulation (TMS) to ameliorate MS spasticity, is still unknown.

Based on these considerations, a prospective and retrospective cohort study of about six years will be performed to assess whether miR-142-3p is a possible biomarker for MS synaptopathy-driven disease progression (AIM1) and for the efficacy of disease-modifying treatments (DMTs) currently used in MS therapy (AIM2a). Moreover, a genetic screening from peripheral blood will be conducted in order to identify single nucleotide polymorphisms (SNPs) in coding and/or regulating regions of miR-142-3p and GLAST/EAAT1 genes, associated with MS synaptopathy (AIM2b). Finally, a repetitive TMS stimulation protocol (iTBS) will be performed in a subgroup of screened MS patients with lower limb spasticity (interventional substudy) to evaluate the patient responsiveness to the treatment linked to the identified SNPs (AIM2c).

Given the heterogeneity and complexity of MS disease, multivariable approach will permit to dissect miR-142-3p contribution to MS course influenced by synaptopathy (AIM1).

Firstly, miR-142-3p levels in MS CSF (the day of recruitment, T0) will be correlated with other possible variables relevant to disease progression, such as:

* clinical (disease duration, estimated as the number of years from onset to the most recent assessment of disability; disability, evaluated using EDSS = Expanded Disability Status Scale; Progression Index, PI = EDSS/disease duration; change in ARR = Annualized Relapse Rate) and neuroradiological parameters (dual-echo proton density; FLAIR = fluid-attenuated inversion recovery; T2-WI = T2-weighted spin-echo images and T1-WI = pre-contrast and post-contrast T1-weighted spin-echo images after intravenous gadolinium (Gd) infusion) at T0 and once per year during a 6-year-follow-up if no relapse occurs (T12, T24, T36, T48, T60 , T72);
* levels of inflammatory and potential excitotoxic protein factors (as IL-1β, TNF and RANTES-CCL5) in the CSF (T0);
* levels of neurofilaments, beta amyloid, tau proteins and growth factors (like NGF, PDGF and BDNF) in the CSF, as possible indicators of neurodegenerative and regenerative processes occurring at the CSF withdrawal (T0).

To reduce the variable dimension, Principal Component Analysis (PCA) will be applied taking into account the contribution of miR-142-3p to disease progression as part of a complex network of molecules circulating in the CSF, and univariable and multivariable correlations will be repeated.

In multivariable analysis (based on multivariable generalized linear models, GLM), miR-142-3p levels in the CSF (or PCA components including miR-142-3p as part of the component) will be considered as the independent variable adjusting for demographical, clinical and neuroradiological values as well as different DMT treatments. A further analysis based on treatment stratifications of the patients will be attempted (AIM2a).

Lastly, the CSF levels of miR-142-3p (or PCA components including miR-142-3p) identified to associate with disease progression variables will be correlated with neurophysiological parameters, recorded by means of TMS to evaluate cortical excitability and plasticity (SICI = short interval intracortical inhibition; ICF = intracortical facilitation; LICI = long interval intracortical inhibition; PAS = Paired Associative Stimulation) in MS patients at T0. Thus, miR-142-3p circulating in the CSF will be validated as possible biomarkers of synaptopathy-driven disease progression (as single molecules or as part of a PCA component).

To identify genetic variants of miR-142-3p and GLAST/EAAT1 coding genes relevant to MS synaptopathy (AIM2b) SNPs will be analyzed at T0 and will be correlated with miR-142-3p levels in the CSF and with other possible variables relevant to disease progression as in AIM1. PCA and GLM models will be applied as in AIM1.

To evaluate treatment responsiveness in the subgroup of screened MS patients included in the interventional substudy based on a two-week protocol of iTBS for reducing lower limb spasticity, the H/M amplitude ratio of the Soleus H reflex and the Modified Ashworth Scale (MAS) will be considered before (W0) and after (W2) the stimulation protocol. Possible association between patient responsiveness to the iTBS stimulation protocol and specific SNPs will be assessed (AIM2c).

Statistical analysis will be performed using Prism GraphPad 6.0, IBM SPSS Statistics 15.0, R software and T-MEV 4.4.1. Data will be tested for normality distribution through the Kolmogorov-Smirnov and Shapiro-Wilk tests. The k-means method will be used to divide MS patients into homogeneous clusters, based on miR-142-3p levels in the CSF and other relevant parameters. Differences between two groups will be analyzed using Student's t-test, Mann-Whitney test, Fisher exact test or log-rank test, as appropriate; multiple comparisons will be performed by ANOVA followed by Tukey HSD or by Kruskal-Wallis. Pearson or nonparametric Spearman correlation coefficients will be performed to evaluate the association of miR-142-3p levels in the CSF or specific genetic variants of MIR142 and SLC1A3 (or the correspondent PCA component, see next) with continuous demographic, clinical and neuroradiological parameters (e.g Age, changes in EDSS, Number of T2 lesions, etc.). For the multiple comparisons it will be controlled the False Discovery Rate (FDR) applying the method proposed by Benjamini and Hochberg.

PCA will be applied to represent sets of potentially correlated variables (CSF levels of miR-142-3p or specific genetic variants of MIR142 and SLC1A3, inflammatory and potential excitotoxic protein factors and levels of neurofilaments, beta amyloid, tau protein and growth factors) with principal components (PC) that are linearly uncorrelated obtained using orthogonal transformation. PCs are ordered so that the first PC has the largest possible variance and only some components are selected to represent the correlated variables. As a result, the dimension of the variables is reduced.

To validate miR-142-3p as biomarker of synaptopathy-driven disease progression (measured in terms of clinical or radiological changes and TMS variables) or specific SNPs of MIR142 and SLC1A3 linked to MS synaptopathy, GLM models will be applied considering, respectively, the miR-142-3p level in the CSF (or the identified PCA components including miRs) or the genetic variants as an independent variable adjusting for demographical, clinical, neuroradiological, neurophysiological, biochemical factors and treatments.

Data will be presented as the mean (standard deviation, sd) or median (25th- 75th percentile). The significance level is established at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent to the study;
* Diagnosis of MS definite according to 2010 revised McDonald's criteria (Polman et al., 2011);
* Age range 18-65 (included);
* EDSS range between 0 and 6 (included);
* Ability to participate to the study protocol.

Exclusion Criteria:

* Inability to provide written informed consent to the study;
* Altered blood count;
* Female with positive pregnancy test at baseline or having active pregnancy plans in the following months after the beginning of the protocol;
* Contraindications to gadolinium (MRI);
* Contraindications to TMS;
* Patients with comorbidities for neurological disease other than MS, included other neurodegenerative chronic diseases or chronic infections (i.e tubercolosis, infectious hepatitis, HIV/AIDS);
* Unstable medical condition or infections;
* Use of medications with increased risk of seizures (i.e. Fampridine, 4- Aminopyridine);
* Concomitant use of drugs that may alter synaptic transmission and plasticity (cannabinoids, L-dopa, antiepiletics, nicotine, baclofen, SSRI, botulinum toxin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
CSF concentration of miR-142-3p | T0 (enrollment); MS patients vs Control subjects
  Quantification of CSF levels of miR-142-3p by qPCR analysis. Relative quantification will be performed by 2^(-ddCt) method.
CSF concentration of soluble molecules | T0 (enrollment); MS patients vs Control subjects
  Quantification of CSF inflammatory molecules (TNF, IL-1β, IL-6, IL-17, IFN-γ, IL1ra, IL-22, IL-2, IL-2ra, IL-10, IL-4, IL-5, IL-13, IL-12p40, IL-8) by Luminex multiplex assays; neurofilaments, beta amyloid, tau proteins and growth factors (like NGF, PDGF and BDNF) by Luminex multiplex assays. Data will be expressed as pg/ml.
Clinical disability assessment by Progression Index calculation for correlation analysis with CSF-miR-142-3p levels | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  Clinical disability will be certified by a qualified neurologist through the Progression Index (PI) calculated as EDSS combined with disease duration (EDSS/disease duration). Disease duration is estimated as the number of years from onset to the most recent assessment of disability and EDSS scale ranging from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Clinical disability assessment by MSFC calculation for correlation analysis with CSF-miR-142-3p levels | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  The Multiple Sclerosis Functional Composite (MSFC) is a three-part composite clinical measure. Three variables were recommended as primary measures: Timed 25-Foot walk; 9-Hole Peg Test; and Paced Auditory Serial Addition Test (PASAT- 3"). The results from each of these three tests are transformed into Z-scores and averaged to yield a composite score for each patient at each time point.
  There are 3 components:
  1. the average scores from the four trials on the 9-HPT;
  2. the average scores of two 25-Foot Timed Walk trials;
  3. the number correct from the PASAT-3. The scores for these three dimensions are combined to create a single score that can be used to detect change over time. This is done by creating Z-scores for each component. MSFC Score = {Zarm, average + Zleg, average + Zcognitive} / 3.0 (Where Zxxx =Z-score) Increased scores represent deterioration in the 9-HPT and the 25-Foot Timed Walk, whereas decreased scores represent deterioration in the PASAT-3.
Neuroradiological assessment for correlation analysis with CSF-miR-142-3p levels | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  By conventional MRI (1.5 Tesla) the following parameters will be evaluated: dual-echo proton density, FLAIR, T1-WI, T2-WI, and contrast-enhanced T1-WI after intravenous gadolinium (Gd) infusion (0.2 ml/kg). A new Gd+ lesion is defined as a typical area of hyperintense signal on postcontrast T1-WI. A new or newly enlarging lesion on T2-WI is defined as a rounded or oval lesion arising from an area previously considered as normal appearing brain tissue and/or showing an identifiable increase in size from a previously stable-appearing lesion. An active scan is defined as showing any new, enlarging or recurrent lesion(s) on postcontrast T1- and T2-WI.
Neurophysiological assessments for correlation analysis with CSF-miR-142-3p levels | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  To assess synaptic excitability by SICI, ICF and LICI, motor thresholds will be calculated at rest as the lowest stimulus intensity able to evoke MEPs of about 50uV in 5 out of 10 consecutive trials (cts), and during a slight voluntary contraction of the target muscle (20-30% of the max voluntary contraction) as the lowest intensity able to evoke MEPs > 100uV in 5 out of 10 cts. The mean peak-to-peak amplitude of the conditioned MEP (cMEP), at each interstimulus interval (ISI), will be expressed as a percentage of the mean peak-to-peak amplitude of the test MEP (tMEP).
  PAS-induced LTP-like plasticity will be expressed as changes of the average MEPs size at each time point after PAS compared to the average baseline MEPs size. Before PAS, 25 MEPs, evoked by single TMS pulses over the APB motor hot spot set at an intensity to obtain MEPs size of about 1mV peak-to-peak, will be collected. The same stimulus intensity will be used to obtain 25 MEPs 0', 30' and 60' after PAS.
Statistical correlation of miR-142-3p levels in MS CSF with disease and neurophysiological parameters | T0 (enrollment), T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months).
  To investigate miR-142-3p association with synaptopathy-driven disease progression (measured in terms of clinical or radiological changes and TMS variables), multivariable generalized linear models (GLM) will be applied considering miR level in the CSF as an independent variable adjusting for demographical, clinical, neuroradiological, neurophysiological, biochemical factors and treatments.
  In the case of unsuccessful identification, Principal Component Analysis (PCA) will be performed to evaluate the miR contribution with other molecules in the CSF (as cytokines, chemokines, growth factors, neurofilaments, beta amyloid and tau protein) to synaptopathy-driven disease progression to reduce the number of variable examined and increase the power of multivariate analysis. Statistical correlations will be repeated on the identified PCA components including miR-142-3p as part of the component. The significance level is established at p<0.05.

SECONDARY OUTCOMES:
Statistical correlation of miR-142-3p levels in MS CSF with patient's responsiveness to disease modifying therapies (DMTs). | Time Frame: T0 (enrollment); Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  miR-142-3p levels in the CSF will be assessed at T0, as reported above. The responsiveness to the DMT, who MS patients underwent as part of their clinical routine, will be evaluated according to clinical and neuroradiological parameters considered in the primary outcomes. Changes in such parameters will be evaluated at different time points during a six-year follow-up (T12-T0; T24-T0, T24-T12, etc). Both univariable and multivariable approaches and stratification of patients based on DMT treatment will be performed.The significance level is established at p<0.05.
Genotyping of SNPs in SLC1A3 and MIR-142 genes for correlation analysis with disease parameters | Time Frame: T0 (enrollment); Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up
  Genetic screening will be performed on peripheral blood withdrawn from MS patients at T0. The following SNPs in MIR142 gene coding for miR-142-3p: rs550842646, rs377637047, rs562696473, rs529802001, rs547987105, rs573562920, rs544684689 and rs549927573, and in SLC1A3 gene coding for GLAST/EAAT1: rs137852620, rs2032892, rs2562582, rs4869675, rs4869676, rs2269272, rs2269273, rs1049522, rs1049524 and rs2731886, will be analyzed.
  Univariable and multivariable correlations of minor allele presence of each screened SNP with clinical, neuroradiological and neurophysiological parameters, detected in the primary outcomes (T0, T12, T24, T36, T48, T60, T72), will allow the identification of SNPs relevant to disease progression. The significance level is established at p<0.05.
Lower limb spasticity assessment by H/M amplitude ratio for the therapeutic TMS substudy | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up; Changes from the starting day (W0) to the end of the 2-week iTBS protocol (W2).
  Lower limb spasticity will be evaluated in all recruited MS patients at T0 and during 6-year-follow-up. A subgroup of MS patients with lower-limb spastic symptoms and carrying SNPs in in SLC1A3 and MIR-142 genes relevant to disease progression will undergo therapeutic iTBS protocol daily for two weeks (interventional substudy) and spasticity will be assessed also immediately before the beginning (W0) and after 2 weeks at the end of the protocol (W2).
  The H/M amplitude ratio of the Soleus H reflex will be evaluated by EMG recordings as an index of spinal excitability. Compound motor action potentials (cMAPs) and H reflex will be evoked by electrical stimulation of the tibial nerve. The maximum amplitudes of the H reflex (H) and CMAP (M) potentials will be measured from peak to peak and H/M ratio was calculated by dividing the maximal amplitude of H wave by that of M wave.
Lower limb spasticity assessment by MAS score for the therapeutic TMS substudy | Changes from T0 (enrollment) to T12 (12 months), T24 (24 months), T36 (36 months), T48 (48 months), T60 (60 months) and T72 (72 months) of follow-up; Changes from the starting day (W0) to the end of the 2-week iTBS protocol (W2).
  Lower limb spasticity will be evaluated in all recruited MS patients at T0 and during 6-year-follow-up. A subgroup of MS patients with lower-limb spastic symptoms and carrying SNPs in in SLC1A3 and MIR-142 genes relevant to disease progression will undergo therapeutic iTBS protocol daily for two weeks (interventional substudy) and spasticity will be assessed also immediately before the beginning (W0) and after 2 weeks at the end of the protocol (W2).
  The Modified Ashworth Scale (MAS) assesses resistance during passive soft-tissue stretching ranging from 0 to 4 score.
Statistical correlation of response to iTBS treatment with MS-significant SNPs of both SLC1A3 and MIR-142. | T0 (enrollment); Changes from the starting day (W0) to the end of the 2-week iTBS protocol (W2).
  Minor allele presence of each screened SNP in SLC1A3 and MIR-142, identified at T0 as relevant to disease progression (see above), will be correlated with changes in spasticity parameters (the H/M amplitude ratio of the Soleus H reflex and MAS score) upon the iTBS treatment (W2-W0). The significance level is established at p<0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — IRCCS Neuromed, Pozzilli, Isernia Italy
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] Mandolesi G, De Vito F, Musella A, Gentile A, Bullitta S, Fresegna D, Sepman H, Di Sanza C, Haji N, Mori F, Buttari F, Perlas E, Ciotti MT, Hornstein E, Bozzoni I, Presutti C, Centonze D. miR-142-3p Is a Key Regulator of IL-1beta-Dependent Synaptopathy in Neuroinflammation. J Neurosci. 2017 Jan 18;37(3):546-561. doi: 10.1523/JNEUROSCI.0851-16.2016. PMID 28100738
- [Background] Mandolesi G, Gentile A, Musella A, Fresegna D, De Vito F, Bullitta S, Sepman H, Marfia GA, Centonze D. Synaptopathy connects inflammation and neurodegeneration in multiple sclerosis. Nat Rev Neurol. 2015 Dec;11(12):711-24. doi: 10.1038/nrneurol.2015.222. Epub 2015 Nov 20. PMID 26585978
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Boffa L, Rimano A, Bernardi G, Koch G, Centonze D. Effects of intermittent theta burst stimulation on spasticity in patients with multiple sclerosis. Eur J Neurol. 2010 Feb;17(2):295-300. doi: 10.1111/j.1468-1331.2009.02806.x. Epub 2009 Oct 23. PMID 19863647
- [Background] Centonze D, Koch G, Versace V, Mori F, Rossi S, Brusa L, Grossi K, Torelli F, Prosperetti C, Cervellino A, Marfia GA, Stanzione P, Marciani MG, Boffa L, Bernardi G. Repetitive transcranial magnetic stimulation of the motor cortex ameliorates spasticity in multiple sclerosis. Neurology. 2007 Mar 27;68(13):1045-50. doi: 10.1212/01.wnl.0000257818.16952.62. PMID 17389310
- [Background] Centonze D, Muzio L, Rossi S, Cavasinni F, De Chiara V, Bergami A, Musella A, D'Amelio M, Cavallucci V, Martorana A, Bergamaschi A, Cencioni MT, Diamantini A, Butti E, Comi G, Bernardi G, Cecconi F, Battistini L, Furlan R, Martino G. Inflammation triggers synaptic alteration and degeneration in experimental autoimmune encephalomyelitis. J Neurosci. 2009 Mar 18;29(11):3442-52. doi: 10.1523/JNEUROSCI.5804-08.2009. PMID 19295150
- [Background] Gandhi R. miRNA in multiple sclerosis: search for novel biomarkers. Mult Scler. 2015 Aug;21(9):1095-103. doi: 10.1177/1352458515578771. Epub 2015 Apr 28. PMID 25921051
- [Background] International Multiple Sclerosis Genetics Consortium; Hafler DA, Compston A, Sawcer S, Lander ES, Daly MJ, De Jager PL, de Bakker PI, Gabriel SB, Mirel DB, Ivinson AJ, Pericak-Vance MA, Gregory SG, Rioux JD, McCauley JL, Haines JL, Barcellos LF, Cree B, Oksenberg JR, Hauser SL. Risk alleles for multiple sclerosis identified by a genomewide study. N Engl J Med. 2007 Aug 30;357(9):851-62. doi: 10.1056/NEJMoa073493. Epub 2007 Jul 29. PMID 17660530
- [Background] Kiselev I, Bashinskaya V, Kulakova O, Baulina N, Popova E, Boyko A, Favorova O. Variants of MicroRNA Genes: Gender-Specific Associations with Multiple Sclerosis Risk and Severity. Int J Mol Sci. 2015 Aug 24;16(8):20067-81. doi: 10.3390/ijms160820067. PMID 26305248
- [Background] Bergman P, Piket E, Khademi M, James T, Brundin L, Olsson T, Piehl F, Jagodic M. Circulating miR-150 in CSF is a novel candidate biomarker for multiple sclerosis. Neurol Neuroimmunol Neuroinflamm. 2016 Apr 20;3(3):e219. doi: 10.1212/NXI.0000000000000219. eCollection 2016 Jun. PMID 27144214
- [Background] Gentile A, Musella A, Bullitta S, Fresegna D, De Vito F, Fantozzi R, Piras E, Gargano F, Borsellino G, Battistini L, Schubart A, Mandolesi G, Centonze D. Siponimod (BAF312) prevents synaptic neurodegeneration in experimental multiple sclerosis. J Neuroinflammation. 2016 Aug 26;13(1):207. doi: 10.1186/s12974-016-0686-4. PMID 27566665
- [Background] Gentile A, Musella A, De Vito F, Fresegna D, Bullitta S, Rizzo FR, Centonze D, Mandolesi G. Laquinimod ameliorates excitotoxic damage by regulating glutamate re-uptake. J Neuroinflammation. 2018 Jan 5;15(1):5. doi: 10.1186/s12974-017-1048-6. PMID 29304807
- [Background] Harris VK, Sadiq SA. Biomarkers of therapeutic response in multiple sclerosis: current status. Mol Diagn Ther. 2014 Dec;18(6):605-17. doi: 10.1007/s40291-014-0117-0. PMID 25164543
- [Background] Housley WJ, Pitt D, Hafler DA. Biomarkers in multiple sclerosis. Clin Immunol. 2015 Nov;161(1):51-8. doi: 10.1016/j.clim.2015.06.015. Epub 2015 Jul 2. PMID 26143623
- [Background] Meinl E, Meister G. MicroRNAs in the CSF: macro-advance in MS? Neurology. 2012 Nov 27;79(22):2162-3. doi: 10.1212/WNL.0b013e31827597d1. Epub 2012 Oct 17. No abstract available. PMID 23077022
- [Background] Quintana E, Ortega FJ, Robles-Cedeno R, Villar ML, Buxo M, Mercader JM, Alvarez-Cermeno JC, Pueyo N, Perkal H, Fernandez-Real JM, Ramio-Torrenta L. miRNAs in cerebrospinal fluid identify patients with MS and specifically those with lipid-specific oligoclonal IgM bands. Mult Scler. 2017 Nov;23(13):1716-1726. doi: 10.1177/1352458516684213. Epub 2017 Jan 9. PMID 28067602
- [Background] Stampanoni Bassi M, Gilio L, Buttari F, Maffei P, Marfia GA, Restivo DA, Centonze D, Iezzi E. Remodeling Functional Connectivity in Multiple Sclerosis: A Challenging Therapeutic Approach. Front Neurosci. 2017 Dec 13;11:710. doi: 10.3389/fnins.2017.00710. eCollection 2017. PMID 29321723